CLINICAL TRIAL: NCT04766970
Title: Telehealth Autism Assessment for Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI resigning from VUMC
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Brianna Lewis, Assistant Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 202427
Record Dates: First submitted 2021-02-11; First posted 2021-02-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized assessment (Active Comparator)
  Interventions: Behavioral: ADOS-2 Module 4
- Telehealth assessment (Experimental)
  Interventions: Behavioral: Adapted Telehealth ADOS-2 Module 4

INTERVENTIONS:
Behavioral: ADOS-2 Module 4 — Assessment in person using standardized Autism Diagnostic Observation Schedule, 2nd Edition (ADOS-2) Module 4.
  Arms: Standardized assessment
Behavioral: Adapted Telehealth ADOS-2 Module 4 — Assessment via telehealth/teleconference platform using an adapted ADOS-2, Module 4 assessment protocol.
  Arms: Telehealth assessment

SUMMARY:
The study aims to investigate the reliability and validity of an adapted Autism Spectrum Disorder assessment measure for use in a telehealth visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* Access to personal computer with video, microphone, and speaker
* English literate
* Fluent English speaker

Exclusion Criteria:

* Non-fluent English speaker
* Not English literate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Concurrent validity | Immediately after intervention
  Concurrent validity will be assessed through correlations between the domain, Overall Total, and calculated Comparison scores of the two ADOS-2 versions, as well as through comparison of total scores on the Social Communication Questionnaire (SCQ) and the Social Responsiveness Scale, Second Edition (SRS-2).

CONTACTS AND LOCATIONS:
Overall Officials: Brianna Lewis, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States